CLINICAL TRIAL: NCT00191698
Title: A Randomized, Double-Blind Comparison of Atomoxetine Hydrochloride and Placebo in Child and Adolescent Outpatients With Attention-Deficit/Hyperactivity Disorder and Comorbid Oppositional Defiant Disorder
Brief Title: Comparison of Atomoxetine and Placebo in Children and Adolescents With ADHD and ODD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7068; B4Z-MC-LYBX
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-10

CONDITIONS: Attention Deficit Hyperactivity Disorder; Oppositional Defiant Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Oppositional Defiant Disorder | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Atomoxetine is administered at 1.2 mg/kg/day, PO for 8 weeks, followed by 1.2 or 2.4 mg/kg/day, PO for 4 weeks, open label administration can continue for up to one year
  Interventions: Drug: atomoxetine hydrochloride
- B (Placebo Comparator): Placebo is administered by mouth, daily for 8 weeks. After 8 weeks, those randomized to placebo may be titrated to 1.2 mg/kg/day atomoxetine for the remainder of the study up to one year
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: atomoxetine hydrochloride
  Other Names: LY139603; Strattera
  Arms: A
Drug: placebo
  Arms: B

SUMMARY:
The purpose of this trial is to test the effectiveness of atomoxetine in treating symptoms of ODD in children with ADHD and ODD.

ELIGIBILITY:
Inclusion Criteria:

* Patients are male or female outpatients who are at least 6 years of age and not more than 12 years of age at study entry.
* Patients must meet DSM-IV diagnostic criteria for ADHD and ODD.
* If other comorbid conditions are present, either the ADHD or the ODD diagnosis must be the patient's primary diagnosis.
* Patients must have laboratory results, including serum chemistries, hematology, and urinalysis showing no significant abnormalities.
* Patients must have an ECG performed at study entry that is absent of any abnormality that, in the opinion of the physician, should exclude the patient.

Exclusion Criteria:

* Patients who weigh less than 20 kg or greater than 60 kg at study entry.
* Patients who have a history of Bipolar I or II disorder, psychosis, or pervasive developmental disorder.
* Patients who have a current diagnosis of Major Depressive Disorder ([MDD]; with or without psychotic features), PTSD, or CDRS-R total raw score >40 at study entry.
* Patients with a history of any seizure disorder.
* Patients determined by the investigator to be at serious suicidal risk.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 226 (Actual)
Dates: Start 2003-12; Primary Completion 2005-06 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Mean reduction in ODD symptoms using the Swanson, Nolan and Pelham Rating Scale-Revised (SNAP-IV), atomoxetine vs placebo | over 8 weeks

SECONDARY OUTCOMES:
Mean change in the investigator-rated SNAP-IV ADHD subscales, atomoxetine vs placebo | over 8 weeks
Mean change in ratings on the Oppositional subscale of the SNAP-IV | over 8 weeks
Mean change in ADHD symptoms by ADHD subscales of the SNAP-IV, 2.4 mg/kg/day vs 1.2 mg/kg/day. | over 4 weeks
Mean change in ratings on the Clinical Global Impressions-Severity (CGI-S). | over 8 weeks
Psychosocial functioning as measured by the total score on the Attention Deficit Hyperactivity Disorder Impact Module (AIM). | over 8 weeks
Environmental stress exacerbation of ODD symptoms by Social Readjustment Rating Scale (SRRS). | 8 weeks, 12 weeks
Adverse events (AEs) | over 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (16):
- Australia (2):
  - For additional information regarding investigative sites for this trial, call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wallsend, New South Wales
  - For additional information regarding investigative sites for this trial, call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parkville, Victoria
- Belgium (3):
  - For additional information regarding investigative sites for this trial, call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Antwerp
  - For additional information regarding investigative sites for this trial, call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
- For additional information regarding investigative sites for this trial, call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Risskov, Denmark
- For additional information regarding investigative sites for this trial, call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Helsinki, Finland
- Germany (2):
  - For additional information regarding investigative sites for this trial, call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mannheim
  - For additional information regarding investigative sites for this trial, call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulm
- Netherlands (2):
  - For additional information regarding investigative sites for this trial, call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nijmegen
  - For additional information regarding investigative sites for this trial, call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Utrecht
- Spain (3):
  - For additional information regarding investigative sites for this trial, call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona, Barcelona
  - For additional information regarding investigative sites for this trial, call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tarrasa, Barcelona
  - For additional information regarding investigative sites for this trial, call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pamplona, Navarre
- United Kingdom (2):
  - For additional information regarding investigative sites for this trial, call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dundee, Augus
  - For additional information regarding investigative sites for this trial, call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edinburgh

REFERENCES:
- [Derived] Bangs ME, Wietecha LA, Wang S, Buchanan AS, Kelsey DK. Meta-analysis of suicide-related behavior or ideation in child, adolescent, and adult patients treated with atomoxetine. J Child Adolesc Psychopharmacol. 2014 Oct;24(8):426-34. doi: 10.1089/cap.2014.0005. Epub 2014 Jul 14. PMID 25019647
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com